CLINICAL TRIAL: NCT07173777
Title: Cardiac Anodal Biphasic Pacing
Acronym: ABP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Rocky Mountain Biphasic (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-46078
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Pacing
Keywords: Anodal biphasic pacing (ABP); Monophasic cathodal pacing (MCP); Ejection fraction; Cardiac implantable electronic device; Cardiac contractility modulation; Implantable cardiac defibrillator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cohort A (Experimental): Cardiac patients who are undergoing interventional cardiac procedure including electrophysiology (EP) with planned retrograde left ventricular access or diagnostic coronary catheterization.
  Interventions: Device: Cardiac Waveform Generator
- Cohort B (Experimental): Patients who have pacing indication and are undergoing routine generator exchange of dual chamber cardiac implantable electronic device (CIED).
  Interventions: Device: Cardiac Waveform Generator
- Cohort C (Experimental): Patients who are undergoing new implant or generator exchange of CIED with cardiac resynchronization therapy.
  Interventions: Device: Cardiac Waveform Generator

INTERVENTIONS:
Device: Cardiac Waveform Generator — A pacing device that allows for programmable pulse waveforms to generate a predefined set of anodal biphasic waveforms. It possesses a battery-powered floating point gate array (FPGA) using software that allows flexibility in waveform configuration.

SUMMARY:
The goal of this study is to test a new pacing method called anodal biphasic pacing (ABP) to determine if this pacing works as well-or better-than current pacing methods. This new method may improve how the heart works and reduce some of the problems caused by regular pacing.

Current implantable pacemakers use a monophasic cathodal waveform to stimulate the heart. Monophasic cathodal pacing (MCP) waveforms slow conduction, impair contractility, cause inflammation, increase risk of atrial fibrillation, heart failure, and mortality. Anodal biphasic pacing (ABP) is an alternative waveform that can stimulate the heart. ABP preconditions the heart and then initiates cardiac contraction. ABP may address the limitations of MCP.

DETAILED DESCRIPTION:
This study is a single-center, prospective, investigator-initiated, non-randomized, study that will investigate ABP in patients with structurally normal hearts and those with non-ischemic cardiomyopathy who are undergoing interventional cardiac procedure, generator exchange of dual chamber Cardiac implantable electronic device (CIED), or de novo implant or generator exchange of CIED with cardiac resynchronization therapy.

Eligible participants, without heart disease and those with nonischemic cardiomyopathy, undergoing CIED implant or generator exchange or interventional cardiac procedure at Boston Medical Center will be screened and prospectively enrolled. Participants will be stratified by left ventricular ejection fraction (EF): those with severely reduced EF (≤35%), mid-range EF (> 35%-49%) and normal EF (EF≥ 50%).

Primary efficacy objectives:

1. To identify which patient populations have the greatest and most consistent hemodynamic benefit from ABP as compared with cathodal pacing.
2. To confirm that ABP does not negatively impact non-responders.
3. To define the ideal anodal biphasic waveform characteristics (amplitude and pulse width) that maximizes the positive effect in subjects who demonstrate hemodynamic improvement ABP
4. To assess differences in capture thresholds between anodal biphasic and cathodal pacing.

Secondary safety objectives:

1. To assess and characterize any ventricular arrhythmias associated with anodal biphasic in comparison to cathodal pacing.
2. To assess device safety
3. To assess procedure safety

ELIGIBILITY:
Inclusion Criteria:

Cohort A

• Planned interventional cardiac procedure

Cohort B

* Planned generator exchange of dual chamber cardiac implantable electronic device (CIED)
* Functioning atrial lead

Cohort C

* Planned de novo implant or generator exchange of CIED with cardiac resynchronization therapy
* Functioning atrial lead

Exclusion Criteria:

* Permanent atrial fibrillation
* Third degree AV block without stable escape rhythm
* Ischemic heart disease or coronary disease > 40%
* Unable to receive heparin
* Are not fluent in English
* Unable to read in English
* Not able to provide informed consent
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Clinically significant maximum rate of pressure change maximum rate of pressure change within the left ventricle during its contraction phase- dP/dtmax. | about 30 minutes
  Response will be expressed as a percent change in these measures with anodal biphasic pacing (ABP) as compared with cathodal pacing. A clinically significant hemodynamic response to pacing will be defined as a >10% increase in dP/dtmax.
Clinically significant stroke work | about 30 minutes
  Response will be expressed as a percent change in these measures with anodal biphasic pacing (ABP) as compared with cathodal pacing. A clinically significant hemodynamic response to pacing will be defined as a >10% increase in stroke work.
Clinically significant left ventricular end-diastolic pressure (LVEDP) | about 30 minutes
  Response will be expressed as a percent change in these measures with anodal biphasic pacing (ABP) as compared with cathodal pacing. A clinically significant hemodynamic response to pacing will be defined as a >10% increase in LVEDP.
Clinically significant diastolic relaxation (tau) | about 30 minutes
  Response will be expressed as a percent change in these measures with anodal biphasic pacing (ABP) as compared with cathodal pacing. A clinically significant hemodynamic response to pacing will be defined as a >10% increase in tau.
Clinically significant volume measurements | about 30 minutes
  Response will be expressed as a percent change in these measures with anodal biphasic pacing (ABP) as compared with cathodal pacing. A clinically significant hemodynamic response to pacing will be defined as a >10% increase in volume measurements.
Capture threshold | about 30 minutes
  This outcome will be measured with decremental pacing threshold testing where pacing output (voltage or pulse width) is decremented until there is a loss of ventricular capture. The minimum output prior to loss of capture is defined as the capture threshold.

SECONDARY OUTCOMES:
Waveform safety concerns | about 30 minutes
  Defined as the development of any of the following with ABP: ventricular tachycardia > 3 beats, premature ventricular contractions at frequency greater than baseline, ventricular couplet, significant drop (>5%) in invasive hemodynamic measures or blood pressure; or any cardioversion for atrial or ventricular arrhythmia.
Device safety issues | about 30 minutes
  Defined as the occurrence of device related adverse event including: device malfunction, failure to output programmed pulse waveform, or failure to output set voltage
Procedural safety issues | about 30 minutes
  Defined as the occurrence of procedure related adverse event including: vascular complication, cardiac complication including cardiac perforation, valvular injury, atrioventricular (AV) or bundle branch block, or thromboembolism.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Helm, MD, Principal Investigator — Boston Medical Center, Cardiology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No